CLINICAL TRIAL: NCT05263791
Title: Evaluating the Non-Inferiority of Airmod to Capnostream™35 on Respiratory Rate Monitoring and User Experience Clinical Evaluation
Brief Title: Evaluating the Non-Inferiority of Airmod to Capnostream™35
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heroic Faith Medical Science Co., Ltd. (Industry)
Collaborators: Elite BioMedical Consulting Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21CT020be
Record Dates: First submitted 2022-01-12; First posted 2022-03-03 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Rate
Keywords: Airmod; Respiratory Rate; Deep learning; Auscultation sound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Airmod (Experimental): The experimental device are installed in the same patient as the reference device to compare the non-inferiority of the respiratory rate measurement.
  Interventions: Device: Airmod

INTERVENTIONS:
Device: Airmod — Both of the respiratory rate monitor (including experimental and reference device) are installed on the enrolled patients. The practitioners can clearly read the result of both devices.

SUMMARY:
This study is a multi-center clinical study of non-invasive medical device in Taiwan. After pre-anaesthesia evaluation, subjects who are suitable for intravenous general anesthesia (IVG) and age 20 years or older will be recruited in this clinical study. 150 subjects will be recruited at this site. The total 300 subjects will be recruited in other clinical centers at En Chu Kong Hospital simultaneously and Cathay General Hospital and Doctor Huang, Chien-Chung of the Anesthesia Department of MacKay Memorial Hospital is the PI of this study. The objective of this study is to evaluate the respiratory rate monitoring performance of "Airmod" respiratory monitoring assistant software, used with the "AccurSound Electronic Stethoscope AS-101" (TFDA Certificate No. 007347) compared to the "Medtronic Capnostream™35 Portable Respiratory Monitor" (TFDA Certificate No. 032283), hereinafter referred to as "comparison method", is non-inferiority than the comparison method. In addition, in order to improve the quality of patient care and ensure safety, this study will also synchronously record the breathing sounds from the " AccurSound Electronic Stethoscope " during the study with the respiratory symptoms of the comparison method, such as: asthma sounds, phlegm sounds, airway infiltration, water accumulation, obstructive sounds, respiratory arrest and respiratory tract edema, and analyze the vital signs for further improvement in the future. Primary Objective: To evaluate accuracy and performance of respiratory rate (RR) measurement from Airmod compared to the comparison method. The primary objective is to establish the non-inferiority. Secondary Objectives: 1. To assess the accuracy of respiratory ate measurement by Airmod comparison with manual-scored auscultation sound during the less sensitive period of Capnography on the comparison method. 2. To measure the agreement between AirRR* and ManCRR*. 3. To evaluate the response time of the first breath detection followed by administration of jaw thrust during the apnea period. The 3rd secondary objective is to compare the response time of Airmod versus the comparison method. 4. To compare the influence of subjects to variated breath rates on respiratory rate monitoring in bpm as measured by Airmod, manual-scored and the Capnostream™35. 5. To evaluate the safety and usability of Airmod. * AirRR Airmod-scored auscultation sound generated from AS-101 * ManCRR Manual-scored Capnography (ManCRR)originated from CapnostreamTM35 (K150272, Medtronic)

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female with at least 20 years of age.
4. Fit for intravenous general anesthesia (IVG) as assessed by pre-anesthesia evaluation.

Exclusion Criteria:

1. Presence of neck pain or injuries.
2. Under the use of high-flow nasal cannula ventilation. Patients with advanced airway management equipment. (For instance, Supraglottic airway device, LMA, Endotracheal tube.) Some equipment, such as High Flow Nasal Cannula (HFNC), CPAP, suction machine, could continually make noise in the patient's airway, affecting auscultation and RR measurement.
3. Unable to wear Airmod and Capnostream™35 device related accessories at the investigator's discretion.
4. As a vulnerable population, including legal incapacity or evidence that a subject cannot understand the purpose and risks of the study, regardless of authorized representative support.
5. Unwilling or unable to comply fully with study procedures (including non-toleration of the capnography cannula) due to any disease condition which can raise doubt about compliance and influencing the study outcome.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - En Chu Kong Hospital, New Taipei City
  - MacKay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atkins JH, Mandel JE. Performance of Masimo rainbow acoustic monitoring for tracking changing respiratory rates under laryngeal mask airway general anesthesia for surgical procedures in the operating room: a prospective observational study. Anesth Analg. 2014 Dec;119(6):1307-14. doi: 10.1213/ANE.0000000000000362. PMID 25025587
- [Background] Hsu FS, Huang SR, Huang CW, Huang CJ, Cheng YR, Chen CC, Hsiao J, Chen CW, Chen LC, Lai YC, Hsu BF, Lin NJ, Tsai WL, Wu YL, Tseng TL, Tseng CT, Chen YT, Lai F. Benchmarking of eight recurrent neural network variants for breath phase and adventitious sound detection on a self-developed open-access lung sound database-HF_Lung_V1. PLoS One. 2021 Jul 1;16(7):e0254134. doi: 10.1371/journal.pone.0254134. eCollection 2021. PMID 34197556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The candidate was invited during their pre-anesthesia appointment and provided with an informed consent form, which explained the details, benefits, and risks of participating in the study. Research staff simultaneously reviewed the candidate's eligibility. The candidate was given at least one day to review and sign the informed consent form before proceeding with the procedures and being formally enrolled in the study.
Groups:
- Airmod: The experimental device are installed in the same patient as the reference device to compare the non-inferiority of the respiratory rate measurement.
  Both of the respiratory rate monitor (including experimental and reference device) are installed on the enrolled patients. The practitioners can clearly read the result of both devices.
  experimenta device: Aimed reference device: "Medtronic Capnostream™35 Portable Respiratory Monitor
Period: Overall Study
Arm/Group | Airmod
Started | 284
Completed | 255
Not Completed | 29

BASELINE CHARACTERISTICS:
Arm/Group | Airmod
Number analyzed (Participants) | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.26 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183
  Male | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 255
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (4.42)
Neck circumference [Mean (Standard Deviation); unit: cm] | 35.74 (4.51)
Height [Mean (Standard Deviation); unit: cm] | 161.81 (7.22)
Weight [Mean (Standard Deviation); unit: kg] | 63.82 (13.44)
Charlson Comorbidity Scale [Count of Participants; unit: Participants] — In the demographic section, the Charlson Comorbidity Index (CCI) was calculated based on the patients' medical history as recorded in their health records, with most conditions being diagnosed by a physician. The index was adjusted for age, assigning 1 point for patients aged 50-59, 2 points for those aged 60-69, 3 points for those aged 70-79, and 4 points for those aged 80 or older. A higher CCI score indicates a worse prognosis and an increased risk of mortality.
  Participants
    0 | 119
    1 | 59
    2 | 36
    3 | 18
    4 | 11
    5 | 7
    6 | 2
    7 | 1
    8 | 1
    9 | 1
American Society of Anesthesiologists' Physical Status Classification [Count of Participants; unit: Participants] — The ASA score was referal to "https://www.asahq.org/standards-and-practice-parameters/statement-on-asa-physical-status-classification-system"
  In brief, ASA I stands for A normal healthy patient, ASA II stands for A patient with mild systemic disease, ASA III stands for A patient with severe systemic disease, ASA IV stands for A patient with severe systemic disease that is a constant threat to life, ASA V stands for A moribund patient who is not expected to survive without the operation, ASA VI stands for A declared brain-dead patient whose organs are being removed for donor purposes.
  Participants
    1 | 17
    2 | 207
    3 | 31

OUTCOME MEASURES:

1. Primary Outcome: Test of the Difference Between airRR and mancRR
Description: The mean difference is based on the comparative pair (reference: mancRR - device under test: airRR) (unit: BPM) The measurement of airRR (airmod recorded breathing rate per minute: BPM ) (minimal: 4 BPM, maximal: 35BPM) The measurement of mancRR (manual scored capnography breathing rate per minute: BPM) (minimal : 0 BPM, maximal 39BPM)
Time Frame: up to 4 hours
Measure: Mean (95% Confidence Interval); unit: breaths per minute
Units Other Than Participants: minute
Arm/Group | Airmod
Number analyzed (Participants) | 255
Number analyzed (minute) | 6920
breaths per minute
  mancRR - airRR | 0.422 [0.3522 to 0.4909]
  airRR | 14.362 [14.2598 to 14.4644]
  mancRR | 14.784 [14.6723 to 14.895]
Statistical Analysis 1: Comparison: Airmod; Hypothesis: airRR-mancRR ≦ -3, In the target of p<0.05 indicates significance; Test type: Non-Inferiority — The primary objective to prove the non-inferiority in between the Airmod and reference device is determined by the difference between AirRR and ManCRR; p < 0.001, Paired t Test

2. Secondary Outcome: Analysis to Assess the Accuracy of Respiratory Rate Measurement by Airmod in Comparison With Manual-scored Auscultation Sound During the Less Sensitive Period of Capnography on Capnostream™35
Description: The mean difference is based on the comparative pair (reference: acoRR - device under test: airRR) (unit: BPM) The measurement of airRR (airmod recorded breathing rate per minute: BPM ) (minimal: 4 BPM, maximal: 35BPM) The measurement of acoRR (manual scored auscultation sound breathing rate per minute: BPM) (minimal : 0 BPM, maximal 60BPM)
Time Frame: up to 4 hours
Measure: Mean (Standard Deviation); unit: breaths per minute
Units Other Than Participants: minute
Arm/Group | Airmod
Number analyzed (Participants) | 255
Number analyzed (minute) | 160
breaths per minute
  airRR | 14.25 (4.15)
  acoRR | 13.14 (5.31)
  airRR-acoRR | 1.11 (3.71)
Statistical Analysis 1: Comparison: Airmod; In this study, a non-inferiority test was conducted during periods of reduced sensitivity in capnography to compare respiratory rate measurements using the Airmod device ("airRR") versus manually scored auscultation sounds (referred to as "acoRR," implying "manARR" in the statistical analysis plan). The research physician identified periods of reduced sensitivity in capnography; Test type: Non-Inferiority — The hypothesis tested is demonstrated airRR non-inferior to acoRR when the capnostream is less sensitive; p < 0.001, Paired t Test

3. Secondary Outcome: Analysis to Measure the Agreement Between AirRR and ManCRR (Limits of Agreement and Bland-Altman Plots)
Description: The Bland-Altman plot and limits of agreement compare the following respiratory rates, all measured in BPM: airRR (Airmod recorded respiratory rate), capRR (capnography recorded respiratory rate), and acoRR (manually scored auscultation respiratory rate) against mancRR (manually scored capnography respiratory rate).
Time Frame: up to 4 hours
Measure: Mean (95% Confidence Interval); unit: breaths per minute
Units Other Than Participants: breaths per minute
Groups:
- Limits of Agreement and Bland-Altman Plots: The experimental device are installed in the same patient as the reference device to compare the non-inferiority of the respiratory rate measurement.
  Airmod: Both of the respiratory rate monitor (including experimental and reference device) are installed on the enrolled patients. The practitioners can clearly read the result of both devices.
Arm/Group | Limits of Agreement and Bland-Altman Plots
Number analyzed (Participants) | 255
Number analyzed (breaths per minute) | 6920
breaths per minute
  manCRR - airRR | 0.42155 [0.3522 to 0.4909]
  manCRR - capRR | -0.0009 [-0.0626 to 0.0608]
  manCRR - acoRR | 0.31701 [0.2506 to 0.3835]

4. Secondary Outcome: Analysis to Evaluate the Response Time of the First Breath Detection Followed by Administration of Jaw Thrust During the Apnea Period
Description: We examined the response time for detecting the first breath after administering a jaw thrust maneuver during an apnea period. The results included the latency of the Airmod breathing response (measured in seconds), the latency of capnography (measured in seconds), and the difference in latency between Airmod and capnography (measured in seconds).
Time Frame: up to 4 hours
Population: In this analysis, we investigated the response time of the first breath detection followed by the administration of a jaw thrust maneuver during the apnea period. As part of the study's third secondary objective, we aimed to compare the response time between the Airmod device and Capnography.
Measure: Mean (Standard Deviation); unit: sec
Units Other Than Participants: event
Arm/Group | Airmod
Number analyzed (Participants) | 255
Number analyzed (event) | 130
sec
  Airmod | 12.61 (14.03)
  Capnography | 28.93 (20.62)
  Airmod-Capnography | -16.32 (21.83)
Statistical Analysis 1: Comparison: Airmod; The hypothesis tested whether the response times obtained with the Airmod device were equal to those recorded with Capnography; Test type: Superiority — This analysis were examined to assess the responsiveness of Airmod and Capnography; p < 0.001, Paired t Test

5. Secondary Outcome: Analysis to Compare the Influence of Subjects to Variated Breath Rates on Respiratory Rate Monitoring in Bpm as Measured by Airmod, Manual-scored and Capnostream™35
Description: as for outcome 1
Time Frame: up to 4 hours
Measure: Mean (95% Confidence Interval); unit: breaths per minute
Units Other Than Participants: breaths per minute
Arm/Group | Airmod
Number analyzed (Participants) | 255
Number analyzed (breaths per minute) | 6920
breaths per minute
  mancRR - airRR | 0.422 [0.3522 to 0.4909]
  airRR | 14.362 [14.2598 to 14.4644]
  mancRR | 14.784 [14.6723 to 14.895]
Statistical Analysis 1: Comparison: Airmod; Hypothesis: airRR-mancRR ≦ -2, In the target of p<0.05 indicates significance; Test type: Non-Inferiority — The objective to prove the non-inferiority in between the Airmod and reference device is determined by the difference between AirRR and ManCRR by subjects; p < 0.05, Paired t Test

6. Secondary Outcome: Safety and Usability of Airmod.
Description: Questionnaire response from research staff, each question score 0 or 1 by candidate, the result stands for successful numbers over all candidates in specific question.
Time Frame: In the study , All participants spend less than 30 min writing thesis questionnaire.
Population: airmod operator
Measure: Number; unit: participants
Groups:
- Airmod Operator: Usability evaluation of airmod
Arm/Group | Airmod Operator
Number analyzed (Participants) | 8
participants
  Were you able to complete this study? (Yes:1, No:0) | 8
  Were you able to turn on Airmod APP? (Yes:1, No:0) | 8
  Were you able to connect Airmod APP to AS-101? (Yes:1, No:0) | 7
  Were you able to record the breath sound ? (Yes:1, No:0) | 8
  Were you able to key in patient's info? (Yes:1, No:0) | 7
  Were you able to adjust the sound playback mode? (Yes:1, No:0) | 8
  Were you able to stop the breath sound recording ? (Yes:1, No:0) | 8
  Were you able to adjust settings? (Yes:1, No:0) | 8
  Were you able to review patient's breath sound recording? (Yes:1, No:0) | 8
  Overall, were you able to use Airmod APP? (Yes:1, No:0) | 8

ADVERSE EVENTS:
Time Frame: up to 4 hours
Arm/Group | Airmod
All-Cause Mortality (participants affected / at risk) | 0/255
Serious Adverse Events (participants affected / at risk) | 0/255
Other Adverse Events (participants affected / at risk) | 0/255

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05263791/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05263791/SAP_001.pdf
  • Informed Consent Form (2021-12-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT05263791/ICF_002.pdf